CLINICAL TRIAL: NCT03569774
Title: The Effect of Individualized PEEP Compared to Low PEEP on Tissue Oxygenation During One Lung Ventilation in Obese Patients Undergoing Thoracic Surgery
Brief Title: Individualized vs Low PEEP in One Lung Ventilation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: Dionne Peacher (Other)
Responsible Party: Sponsor-Investigator, Dionne Peacher, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201805831
Record Dates: First submitted 2018-06-02; First posted 2018-06-26 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: One-Lung Ventilation; Obesity; Lung Diseases
MeSH Terms: conditions — Obesity; Lung Diseases | interventions — One-Lung Ventilation

STUDY DESIGN:
Intervention Model Description: Mechanical ventilation with individualized PEEP will be compared to mechanical ventilating with low PEEP during lung isolation in each subject. Each subject will receive one PEEP level then will receive the second PEEP level. The order in which each subject receives the PEEP level will be randomized.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized PEEP (Experimental): Individualized PEEP will be identified by performing a decremental PEEP protocol which will determine the level of PEEP that correlates with maximal lung compliance in each subject. Subjects will receive one-lung ventilation with individualized PEEP
  Interventions: Procedure: One-lung ventilation with individualized PEEP
- Low PEEP (Active Comparator): Subjects will receive One-lung ventilation with low PEEP (5 cmH2O)
  Interventions: Procedure: One-lung ventilation with low PEEP

INTERVENTIONS:
Procedure: One-lung ventilation with individualized PEEP — During one-lung ventilation for lung resection surgery, PEEP will be applied. After a subject's individualized PEEP (PEEP that corresponds to maximum lung compliance) is determined, the subject will receive one-lung ventilation with individualized PEEP.
  Arms: Individualized PEEP
Procedure: One-lung ventilation with low PEEP — Subjects will receive one-lung ventilation with low PEEP (5 cmH2O)
  Arms: Low PEEP

SUMMARY:
The aim of the prospective crossover study is to investigate the effect of individualized positive end-expiratory pressure (PEEP) on measures of tissue oxygenation, compared with low PEEP.

DETAILED DESCRIPTION:
During surgery on the lung, ventilation of one lung at a time is often necessary. During thoracic surgery requiring one-lung ventilation (OLV), hypoxemia (reduced oxygen tension in blood) can present a clinical challenge. Due to multiple factors, the likelihood of hypoxemia during OLV in obese patients is increased. Atelectasis (collapse of the lung airspaces) contributes to hypoxemia and can be mitigated by application of recruitment maneuvers and positive end-expiratory pressure (PEEP). A recruitment maneuver is a breath given in a mechanically ventilated patient that helps to open up collapsed air spaces, and PEEP is application of a continuous amount of positive pressure that helps keep the air spaces open at the end of an exhaled breath. Adjusting the level of PEEP to each individual patient's optimal lung compliance (individualized PEEP) improves blood oxygen levels compared to application of standard low PEEP (5 cmH2O); however, higher levels of PEEP required to achieve optimal lung compliance could increase intrathoracic pressures to a level that impedes normal circulation. This could negatively affect blood flow (cardiac output) and delivery of oxgyen to vital organs.

Evidence addressing OLV in obese patients is lacking. The purpose of this study is to compare brain oxygen levels (cerebral oxygen saturation) and measures of blood flow and gas exchange during OLV with individualized PEEP vs low standard PEEP in obese patients undergoing thoracic surgery. To our knowledge, there is no previous study that compares oxygen delivery to vital organs (such as the brain) during OLV using individualized PEEP versus standard low PEEP, in an obese patient population.

In this study, subjects undergoing OLV during surgery to remove a portion of the lung (lobectomy) will undergo a process to determine their individualized PEEP and then two 20-minute experimental periods-- one period with OLV with low PEEP and one period with OLV with individualized PEEP. Measurements of cerebral oxygen saturation, blood oxygen levels, cardiac output, and blood pressure medication dose will be measuring before and after these experimental periods during surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject undergoing elective pulmonary lobectomy requiring one-lung ventilation
2. Body-mass index ≥ 30 kg/m2
3. Age ≥ 18 years and ≤ 80 years

Exclusion Criteria:

1. Age ≤ 18 year or ≥ 80 years
2. Moderate or severe cardiac valvular disease
3. Left ventricular ejection fraction < 30%
4. Moderate or severe right ventricular systolic dysfunction
5. Severe pulmonary hypertension
6. Presence of pulmonary bullae or blebs on preoperative chest imaging studies (e.g., radiograph, computed tomograph)
7. Emergency surgery
8. Previous history of lung surgery on the non-operative lung
9. Pregnancy
10. Incarceration
11. Mental incapacitation
12. Patient refusal
13. Non-English speaking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Cerebral oximetry | Change from baseline cerebral oximetry at the end of each intraoperative 20 minute experimental period. All measurements are made during the 4-6 hour surgery.
  Cerebral oximetry (a measure of oxygen levels in the brain) as measured by near-infrared spectroscopy (noninvasive monitor applied to the forehead)

SECONDARY OUTCOMES:
Arterial blood oxygen tension (PaO2) | Measured at baseline, and then at the end of each 20 minute intraoperative experimental period. All measurements are made during the 4-6 hour surgery.
  A measure of oxygen level in arterial blood
Venous blood oxygen tension (PvO2) | Measured at baseline, and then at the end of each 20 minute intraoperative experimental period. All measurements are made during the 4-6 hour surgery.
  A measure of oxygen level in venous blood
Venous blood oxygen saturation (SvO2) | Measured at baseline, and then at the end of each 20 minute intraoperative experimental period. All measurements are made during the 4-6 hour surgery.
  A measure of oxygen saturation in venous blood
Cardiac output | Measured at baseline, and then at the end of each 20 minute intraoperative experimental period. All measurements are made during the 4-6 hour surgery.
  A measure of blood flow throughout the body
Phenylephrine dose | Total dose of phenylephrine administered during each intraoperative 20 minute experimental period. All measurements are made during the 4-6 hour surgery.
  Total dose of phenylephrine (medication used to raise blood pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Dionne Peacher, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal

REFERENCES:
- [Background] Campos JH, Feider A. Hypoxia During One-Lung Ventilation-A Review and Update. J Cardiothorac Vasc Anesth. 2018 Oct;32(5):2330-2338. doi: 10.1053/j.jvca.2017.12.026. Epub 2017 Dec 19. No abstract available. PMID 29361458
- [Background] Karzai W, Schwarzkopf K. Hypoxemia during one-lung ventilation: prediction, prevention, and treatment. Anesthesiology. 2009 Jun;110(6):1402-11. doi: 10.1097/ALN.0b013e31819fb15d. PMID 19417615
- [Background] Ferrando C, Mugarra A, Gutierrez A, Carbonell JA, Garcia M, Soro M, Tusman G, Belda FJ. Setting individualized positive end-expiratory pressure level with a positive end-expiratory pressure decrement trial after a recruitment maneuver improves oxygenation and lung mechanics during one-lung ventilation. Anesth Analg. 2014 Mar;118(3):657-65. doi: 10.1213/ANE.0000000000000105. PMID 24557111
- [Background] de Matos GF, Stanzani F, Passos RH, Fontana MF, Albaladejo R, Caserta RE, Santos DC, Borges JB, Amato MB, Barbas CS. How large is the lung recruitability in early acute respiratory distress syndrome: a prospective case series of patients monitored by computed tomography. Crit Care. 2012 Jan 8;16(1):R4. doi: 10.1186/cc10602. PMID 22226331
- [Background] Borges JB, Okamoto VN, Matos GF, Caramez MP, Arantes PR, Barros F, Souza CE, Victorino JA, Kacmarek RM, Barbas CS, Carvalho CR, Amato MB. Reversibility of lung collapse and hypoxemia in early acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Aug 1;174(3):268-78. doi: 10.1164/rccm.200506-976OC. Epub 2006 May 11. PMID 16690982
- [Background] Writing Group for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART) Investigators; Cavalcanti AB, Suzumura EA, Laranjeira LN, Paisani DM, Damiani LP, Guimaraes HP, Romano ER, Regenga MM, Taniguchi LNT, Teixeira C, Pinheiro de Oliveira R, Machado FR, Diaz-Quijano FA, Filho MSA, Maia IS, Caser EB, Filho WO, Borges MC, Martins PA, Matsui M, Ospina-Tascon GA, Giancursi TS, Giraldo-Ramirez ND, Vieira SRR, Assef MDGPL, Hasan MS, Szczeklik W, Rios F, Amato MBP, Berwanger O, Ribeiro de Carvalho CR. Effect of Lung Recruitment and Titrated Positive End-Expiratory Pressure (PEEP) vs Low PEEP on Mortality in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1335-1345. doi: 10.1001/jama.2017.14171. PMID 28973363